CLINICAL TRIAL: NCT02741180
Title: Sparsity-based Magnetic Resonance Imaging of Cardiac Arrhythmias
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-00116
Record Dates: First submitted 2016-03-29; First posted 2016-04-18 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrythmias
MeSH Terms: interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Arrhythmias (Other)
  Interventions: Other: 3D Imaging; Other: Late Gadolinium Enhancement (LGE)
- Healthy Control (Other)
  Interventions: Other: 3D Imaging; Other: Late Gadolinium Enhancement (LGE)

INTERVENTIONS:
Other: 3D Imaging — "roadmapping" of electrophysiology (EP) procedures
Other: Late Gadolinium Enhancement (LGE) — useful for delineating abnormal myocardium, including fibrotic regions that can serve as sources of arrhythmias.

SUMMARY:
The primary purpose of this study is to improve the quality of Magnetic Resonance Imaging in patients with heart arrhythmia. Investigators will recruit 105 patients with arrhythmia and 30 control volunteers over 3 years and will use two arrhythmia-tolerant imaging methods for diagnosis.

DETAILED DESCRIPTION:
In the proposed research, investigators will extend conventional cardiac magnetic resonance methods to enable the creation of high-quality cine CMR images in the presence of multiple kinds of arrhythmia. Two arrhythmia-tolerant imaging methods will be adopted, which are particularly useful in arrhythmia: 1) 3D imaging, which is useful for many purposes, including "road mapping" of electrophysiology (EP) procedures, and 2) late gadolinium enhancement (LGE), which is useful for delineating abnormal myocardium, including fibrotic regions that can serve as sources of arrhythmias.

ELIGIBILITY:
Inclusion Criteria for Arrhythmia Patients:

* Patients diagnosed with heart arrhythmia scheduled for routine clinical MRI examinations).
* Patients scheduled for routine clinical MRI examinations who do not have a specific known diagnosis of arrhythmia, but who may be found to have image degradation due to arrhythmia during the CMR examination.

Inclusion Criteria for Controls:

* No history of heart arrhythmia.

Exclusion Criteria for Patients and Controls:

* Hemodynamic instability.
* Contraindications for MRI examinations (e.g., pacemakers or ferromagnetic vascular clips).
* History of prior cardiovascular disease or significant risk factors:

  * Diabetes, hypertension, smoking, and hyperlipidemia, etc.

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Paired-sample Wilcoxon signed rank test to evaluate measures on Likert scales | 3 Years
Paired-sample t tests for quantitative measures of intensity of image artifacts | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Leon Axel, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States